CLINICAL TRIAL: NCT03412838
Title: Factors Influencing Bone Block Allograft Resorption. A Randomized Clinical Trial
Brief Title: Factors Influencing Bone Block Allograft Resorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Associate Profesor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-15/566
Record Dates: First submitted 2018-01-14; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Graft Loss
Keywords: Bone block allograft; Bone density; Graft resorption; PRP; RCT

STUDY DESIGN:
Intervention Model Description: Twenty-eight patients referred for implant placement and with insufficient bucco-lingual (BL) alveolar bone width (<4 mm) were included in the study. Patients received freeze dried bone allograft (FDBA) blocks of either allogeneic cancellous or cortico-cancellous bone obtained from the iliac crest. Patients included in the clinical trial were randomly allocated by a blinded assistant in two groups: in the cortico-cancellous group (CC), and cancellous group (C).
Who Masked: Participant, Investigator
Masking Description: Patients included in the clinical trial were randomly allocated by a blinded assistant in two groups: in the cortico-cancellous group (CC), and cancellous group (C). Allocation of participants to intervention groups in a truly unpredictable, randomized sequence was performed using a computerized random number generated by the GraphPadQuickCalc software (GraphPad Software Inc., La Jolla, CA). Blocked randomization was performed to maintain equal group size. As a result 14 patients were randomly assigned to de CC group and other 14 to the C group. All bone augmentation surgeries were performed by the same oral surgeon, with expertise on block surgeries (JT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cortico-Cancellous (Active Comparator): Graft surgery with cortico-cancellous block, freeze dried bone allograft (FDBA) for treatment the atrophic maxilla prior implant placement
  Interventions: Procedure: graft surgery
- Cancellous (Active Comparator): Graft surgery with cancellous block, freeze dried bone allograft (FDBA) for treatment the atrophic maxilla prior implant placement
  Interventions: Procedure: graft surgery

INTERVENTIONS:
Procedure: graft surgery — A graft surgery using bone allogenic blocks that are screwed over the atrophic sites of the maxilla to obtain bone augmentation to support dental implants

SUMMARY:
A main drawback of bone block graft surgery is the resorption occurring in early stages of healing. The aim of this work was investigate different factors associated with graft resorption in allogeneic bone block graft surgery.

DETAILED DESCRIPTION:
Introduction: A main drawback of bone block graft surgery is the resorption occurring in early stages of healing. The aim of this work was investigate different factors associated with graft resorption in allogeneic bone block graft surgery.

Materials and methods: Twenty-eight patients referred for implant placement and with insufficient bucco-lingual (BL) alveolar bone width (<4 mm) were included in the study. Patients received freeze dried bone allograft (FDBA) blocks of either allogeneic cancellous or cortico-cancellous bone obtained from the iliac crest. The aforementioned groups were compared in regards to bone resorption using General Estimating Equations (GEE) and logistic regression. Demographic data, trabecular bone density, graft site were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Twenty eight totally and partially edentulous patients referred for dental implant therapy from January 2011 to September 2015 were enrolled in the study. All patients had insufficient bucco-lingual (BL) alveolar bone width (<4 mm) that prevented placement of regular size implants

Exclusion Criteria:

* Patients with severe systemic disease (American Society of Anesthesiology III or IV) were excluded from the study. In addition, patients who were pregnant, or patients with diseases affecting bone, such as Paget's disease, osteomalacia, diabetes, vitamin D deficiency, alcoholism, hyperthyroidism cancer or osteoporosis as well as those on medications that might affect bone metabolism, such as bisphosphonates, corticosteroids or antiepileptic medicaments were also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Bone Augmentation | 0 months
  A region of interest (ROI) containing the entire trabecular bone area of the alveolar ridge was created using the closed polygon tool of the OsiriX software.

SECONDARY OUTCOMES:
Percentage of bone resorption | 4 months
  A region of interest (ROI) containing the entire trabecular bone area of the alveolar ridge was created using the closed polygon tool of the OsiriX software.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Torres, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu JH, Wang HL. Horizontal bone augmentation: the decision tree. Int J Periodontics Restorative Dent. 2011 Jul-Aug;31(4):429-36. PMID 21837309
- [Background] Nevins M, Mellonig JT. The advantages of localized ridge augmentation prior to implant placement: a staged event. Int J Periodontics Restorative Dent. 1994 Apr;14(2):96-111. PMID 7928133
- [Background] Lundgren S, Sjostrom M, Nystrom E, Sennerby L. Strategies in reconstruction of the atrophic maxilla with autogenous bone grafts and endosseous implants. Periodontol 2000. 2008;47:143-61. doi: 10.1111/j.1600-0757.2008.00265.x. No abstract available. PMID 18412579
- [Background] Grunder U, Gracis S, Capelli M. Influence of the 3-D bone-to-implant relationship on esthetics. Int J Periodontics Restorative Dent. 2005 Apr;25(2):113-9. PMID 15839587
- [Background] Misch CM. Comparison of intraoral donor sites for onlay grafting prior to implant placement. Int J Oral Maxillofac Implants. 1997 Nov-Dec;12(6):767-76. PMID 9425757
- [Background] McAllister BS, Haghighat K. Bone augmentation techniques. J Periodontol. 2007 Mar;78(3):377-96. doi: 10.1902/jop.2007.060048. PMID 17335361
- [Background] Zmolek JC, Dorr LD. Revision total hip arthroplasty. The use of solid allograft. J Arthroplasty. 1993 Aug;8(4):361-70. doi: 10.1016/s0883-5403(06)80034-3. PMID 8409987
- [Background] Haddad FS, Spangehl MJ, Masri BA, Garbuz DS, Duncan CP. Circumferential allograft replacement of the proximal femur. A critical analysis. Clin Orthop Relat Res. 2000 Feb;(371):98-107. doi: 10.1097/00003086-200002000-00011. PMID 10693554
- [Background] Chiapasco M, Colletti G, Coggiola A, Di Martino G, Anello T, Romeo E. Clinical outcome of the use of fresh frozen allogeneic bone grafts for the reconstruction of severely resorbed alveolar ridges: preliminary results of a prospective study. Int J Oral Maxillofac Implants. 2015 Mar-Apr;30(2):450-60. doi: 10.11607/jomi.3763. PMID 25830406
- [Background] Barone A, Varanini P, Orlando B, Tonelli P, Covani U. Deep-frozen allogeneic onlay bone grafts for reconstruction of atrophic maxillary alveolar ridges: a preliminary study. J Oral Maxillofac Surg. 2009 Jun;67(6):1300-6. doi: 10.1016/j.joms.2008.12.043. PMID 19446220
- [Background] Peleg M, Sawatari Y, Marx RN, Santoro J, Cohen J, Bejarano P, Malinin T. Use of corticocancellous allogeneic bone blocks for augmentation of alveolar bone defects. Int J Oral Maxillofac Implants. 2010 Jan-Feb;25(1):153-62. PMID 20209198
- [Background] Waasdorp J, Reynolds MA. Allogeneic bone onlay grafts for alveolar ridge augmentation: a systematic review. Int J Oral Maxillofac Implants. 2010 May-Jun;25(3):525-31. PMID 20556251
- [Background] Ehrler DM, Vaccaro AR. The use of allograft bone in lumbar spine surgery. Clin Orthop Relat Res. 2000 Feb;(371):38-45. doi: 10.1097/00003086-200002000-00005. PMID 10693548
- [Background] Contar CM, Sarot JR, Bordini J Jr, Galvao GH, Nicolau GV, Machado MA. Maxillary ridge augmentation with fresh-frozen bone allografts. J Oral Maxillofac Surg. 2009 Jun;67(6):1280-5. doi: 10.1016/j.joms.2008.11.010. PMID 19446217
- [Background] Acocella A, Bertolai R, Ellis E 3rd, Nissan J, Sacco R. Maxillary alveolar ridge reconstruction with monocortical fresh-frozen bone blocks: a clinical, histological and histomorphometric study. J Craniomaxillofac Surg. 2012 Sep;40(6):525-33. doi: 10.1016/j.jcms.2011.09.004. Epub 2011 Nov 9. PMID 22075326
- [Background] Carinci F, Brunelli G, Franco M, Viscioni A, Rigo L, Guidi R, Strohmenger L. A retrospective study on 287 implants installed in resorbed maxillae grafted with fresh frozen allogenous bone. Clin Implant Dent Relat Res. 2010 Jun 1;12(2):91-8. doi: 10.1111/j.1708-8208.2008.00133.x. Epub 2008 Dec 3. PMID 19076178
- [Background] Nissan J, Marilena V, Gross O, Mardinger O, Chaushu G. Histomorphometric analysis following augmentation of the anterior atrophic maxilla with cancellous bone block allograft. Int J Oral Maxillofac Implants. 2012 Jan-Feb;27(1):84-9. PMID 22299083
- [Background] Al-Abedalla K, Torres J, Cortes AR, Wu X, Nader SA, Daniel N, Tamimi F. Bone Augmented With Allograft Onlays for Implant Placement Could Be Comparable With Native Bone. J Oral Maxillofac Surg. 2015 Nov;73(11):2108-22. doi: 10.1016/j.joms.2015.06.151. Epub 2015 Jun 20. PMID 26126920
- [Background] Lumetti S, Consolo U, Galli C, Multinu A, Piersanti L, Bellini P, Manfredi E, Corinaldesi G, Zaffe D, Macaluso GM, Marchetti C. Fresh-frozen bone blocks for horizontal ridge augmentation in the upper maxilla: 6-month outcomes of a randomized controlled trial. Clin Implant Dent Relat Res. 2014 Feb;16(1):116-23. doi: 10.1111/j.1708-8208.2012.00458.x. Epub 2012 Apr 24. PMID 22530793
- [Background] Lumetti S, Galli C, Manfredi E, Consolo U, Marchetti C, Ghiacci G, Toffoli A, Bonanini M, Salgarelli A, Macaluso GM. Correlation between density and resorption of fresh-frozen and autogenous bone grafts. Biomed Res Int. 2014;2014:508328. doi: 10.1155/2014/508328. Epub 2014 Jun 24. PMID 25050354
- [Background] Chiapasco M, Di Martino G, Anello T, Zaniboni M, Romeo E. Fresh frozen versus autogenous iliac bone for the rehabilitation of the extremely atrophic maxilla with onlay grafts and endosseous implants: preliminary results of a prospective comparative study. Clin Implant Dent Relat Res. 2015 Jan;17 Suppl 1:e251-66. doi: 10.1111/cid.12191. Epub 2013 Dec 27. PMID 24373321
- [Background] Spin-Neto R, Landazuri Del Barrio RA, Pereira LA, Marcantonio RA, Marcantonio E, Marcantonio E Jr. Clinical similarities and histological diversity comparing fresh frozen onlay bone blocks allografts and autografts in human maxillary reconstruction. Clin Implant Dent Relat Res. 2013 Aug;15(4):490-7. doi: 10.1111/j.1708-8208.2011.00382.x. Epub 2011 Aug 11. PMID 21834864
- [Background] Spin-Neto R, Stavropoulos A, Coletti FL, Faeda RS, Pereira LA, Marcantonio E Jr. Graft incorporation and implant osseointegration following the use of autologous and fresh-frozen allogeneic block bone grafts for lateral ridge augmentation. Clin Oral Implants Res. 2014 Feb;25(2):226-33. doi: 10.1111/clr.12107. Epub 2013 Jan 25. PMID 23346871
- [Background] Donovan MG, Dickerson NC, Hellstein JW, Hanson LJ. Autologous calvarial and iliac onlay bone grafts in miniature swine. J Oral Maxillofac Surg. 1993 Aug;51(8):898-903. doi: 10.1016/s0278-2391(10)80112-0. PMID 8336227
- [Background] Anitua E. Plasma rich in growth factors: preliminary results of use in the preparation of future sites for implants. Int J Oral Maxillofac Implants. 1999 Jul-Aug;14(4):529-35. PMID 10453668
- [Background] Alonso N, Machado de Almeida O, Jorgetti V, Amarante MT. Cranial versus iliac onlay bone grafts in the facial skeleton: a macroscopic and histomorphometric study. J Craniofac Surg. 1995 Mar;6(2):113-8; discussion 119. doi: 10.1097/00001665-199503000-00006. PMID 8601015
- [Background] Zins JE, Whitaker LA. Membranous versus endochondral bone: implications for craniofacial reconstruction. Plast Reconstr Surg. 1983 Dec;72(6):778-85. doi: 10.1097/00006534-198312000-00005. PMID 6196801
- [Background] Hardesty RA, Marsh JL. Craniofacial onlay bone grafting: a prospective evaluation of graft morphology, orientation, and embryonic origin. Plast Reconstr Surg. 1990 Jan;85(1):5-14; discussion 15. PMID 2293737
- [Background] Ozaki W, Buchman SR. Volume maintenance of onlay bone grafts in the craniofacial skeleton: micro-architecture versus embryologic origin. Plast Reconstr Surg. 1998 Aug;102(2):291-9. doi: 10.1097/00006534-199808000-00001. PMID 9703062
- [Background] Ozaki W, Buchman SR, Goldstein SA, Fyhrie DP. A comparative analysis of the microarchitecture of cortical membranous and cortical endochondral onlay bone grafts in the craniofacial skeleton. Plast Reconstr Surg. 1999 Jul;104(1):139-47. PMID 10597686
- [Background] Buffoli B, Boninsegna R, Rezzani R, Poli PP, Santoro F, Rodella LF. Histomorphometrical evaluation of fresh frozen bone allografts for alveolar bone reconstruction: preliminary cases comparing femoral head with iliac crest grafts. Clin Implant Dent Relat Res. 2013 Dec;15(6):791-8. doi: 10.1111/cid.12028. Epub 2013 Jan 7. PMID 23294489
- [Background] Keith JD Jr, Petrungaro P, Leonetti JA, Elwell CW, Zeren KJ, Caputo C, Nikitakis NG, Schopf C, Warner MM. Clinical and histologic evaluation of a mineralized block allograft: results from the developmental period (2001-2004). Int J Periodontics Restorative Dent. 2006 Aug;26(4):321-7. PMID 16939013
- [Background] Chiapasco M, Autelitano L, Rabbiosi D, Zaniboni M. The role of pericranium grafts in the reduction of postoperative dehiscences and bone resorption after reconstruction of severely deficient edentulous ridges with autogenous onlay bone grafts. Clin Oral Implants Res. 2013 Jun;24(6):679-87. doi: 10.1111/j.1600-0501.2012.02485.x. Epub 2012 May 3. PMID 22551410
- [Background] Nissan J, Marilena V, Gross O, Mardinger O, Chaushu G. Histomorphometric analysis following augmentation of the posterior mandible using cancellous bone-block allograft. J Biomed Mater Res A. 2011 Jun 15;97(4):509-13. doi: 10.1002/jbm.a.33096. Epub 2011 Apr 20. PMID 21509934
- [Background] Norton MR, Gamble C. Bone classification: an objective scale of bone density using the computerized tomography scan. Clin Oral Implants Res. 2001 Feb;12(1):79-84. doi: 10.1034/j.1600-0501.2001.012001079.x. PMID 11168274
- [Background] Jaffin RA, Berman CL. The excessive loss of Branemark fixtures in type IV bone: a 5-year analysis. J Periodontol. 1991 Jan;62(1):2-4. doi: 10.1902/jop.1991.62.1.2. PMID 2002427
- [Background] Esposito M, Hirsch JM, Lekholm U, Thomsen P. Biological factors contributing to failures of osseointegrated oral implants. (I). Success criteria and epidemiology. Eur J Oral Sci. 1998 Feb;106(1):527-51. doi: 10.1046/j.0909-8836..t01-2-.x. PMID 9527353
- [Background] He YX, Zhang G, Pan XH, Liu Z, Zheng LZ, Chan CW, Lee KM, Cao YP, Li G, Wei L, Hung LK, Leung KS, Qin L. Impaired bone healing pattern in mice with ovariectomy-induced osteoporosis: A drill-hole defect model. Bone. 2011 Jun 1;48(6):1388-400. doi: 10.1016/j.bone.2011.03.720. Epub 2011 Mar 21. PMID 21421090
- [Background] Foger-Samwald U, Patsch JM, Schamall D, Alaghebandan A, Deutschmann J, Salem S, Mousavi M, Pietschmann P. Molecular evidence of osteoblast dysfunction in elderly men with osteoporotic hip fractures. Exp Gerontol. 2014 Sep;57:114-21. doi: 10.1016/j.exger.2014.05.014. Epub 2014 May 24. PMID 24862290
- [Background] Foger-Samwald U, Vekszler G, Horz-Schuch E, Salem S, Wipperich M, Ritschl P, Mousavi M, Pietschmann P. Molecular mechanisms of osteoporotic hip fractures in elderly women. Exp Gerontol. 2016 Jan;73:49-58. doi: 10.1016/j.exger.2015.11.012. Epub 2015 Dec 1. PMID 26608808
- [Background] Levin L, Kessler-Baruch O. Cigarette smoking and the alveolar bone around teeth and dental implants. N Y State Dent J. 2013 Aug-Sep;79(5):53-9. PMID 24245464
- [Background] Belser UC, Schmid B, Higginbottom F, Buser D. Outcome analysis of implant restorations located in the anterior maxilla: a review of the recent literature. Int J Oral Maxillofac Implants. 2004;19 Suppl:30-42. PMID 15635944
- [Background] Torres J, Tamimi F, Martinez PP, Alkhraisat MH, Linares R, Hernandez G, Torres-Macho J, Lopez-Cabarcos E. Effect of platelet-rich plasma on sinus lifting: a randomized-controlled clinical trial. J Clin Periodontol. 2009 Aug;36(8):677-87. doi: 10.1111/j.1600-051X.2009.01437.x. Epub 2009 Jun 26. PMID 19563329
- [Background] Chaushu G, Mardinger O, Peleg M, Ghelfan O, Nissan J. Analysis of complications following augmentation with cancellous block allografts. J Periodontol. 2010 Dec;81(12):1759-64. doi: 10.1902/jop.2010.100235. Epub 2010 Aug 3. PMID 20681816
- [Background] Torres J, Tamimi F, Alkhraisat MH, Manchon A, Linares R, Prados-Frutos JC, Hernandez G, Lopez Cabarcos E. Platelet-rich plasma may prevent titanium-mesh exposure in alveolar ridge augmentation with anorganic bovine bone. J Clin Periodontol. 2010 Oct;37(10):943-51. doi: 10.1111/j.1600-051X.2010.01615.x. PMID 20796106
- [Background] Bouletreau PJ, Warren SM, Spector JA, Peled ZM, Gerrets RP, Greenwald JA, Longaker MT. Hypoxia and VEGF up-regulate BMP-2 mRNA and protein expression in microvascular endothelial cells: implications for fracture healing. Plast Reconstr Surg. 2002 Jun;109(7):2384-97. doi: 10.1097/00006534-200206000-00033. PMID 12045566
- [Background] Ishida K, Matsumoto T, Sasaki K, Mifune Y, Tei K, Kubo S, Matsushita T, Takayama K, Akisue T, Tabata Y, Kurosaka M, Kuroda R. Bone regeneration properties of granulocyte colony-stimulating factor via neovascularization and osteogenesis. Tissue Eng Part A. 2010 Oct;16(10):3271-84. doi: 10.1089/ten.tea.2009.0268. PMID 20626235
- [Background] Nahles S, Nack C, Gratecap K, Lage H, Nelson JJ, Nelson K. Bone physiology in human grafted and non-grafted extraction sockets--an immunohistochemical study. Clin Oral Implants Res. 2013 Jul;24(7):812-9. doi: 10.1111/j.1600-0501.2012.02462.x. Epub 2012 Mar 30. PMID 22462496
- [Background] Alleyne B, Varghai D, Askeroglu U, Zwiebel S, Tobin K, Gosain AK. The Impact of Age Upon Healing: Absolute Quantification of Osteogenic Genes in Calvarial Critical-Sized Defects. J Craniofac Surg. 2016 Jan;27(1):258-63. doi: 10.1097/SCS.0000000000001313. PMID 26751427
- [Background] Viscioni A, Franco M, Rigo L, Guidi R, Spinelli G, Carinci F. Retrospective study of standard-diameter implants inserted into allografts. J Oral Maxillofac Surg. 2009 Feb;67(2):387-93. doi: 10.1016/j.joms.2008.06.099. PMID 19138615
- [Background] Nissan J, Ghelfan O, Mardinger O, Calderon S, Chaushu G. Efficacy of cancellous block allograft augmentation prior to implant placement in the posterior atrophic mandible. Clin Implant Dent Relat Res. 2011 Dec;13(4):279-85. doi: 10.1111/j.1708-8208.2009.00219.x. Epub 2009 Aug 5. PMID 19673921
- [Background] Nissan J, Mardinger O, Calderon S, Romanos GE, Chaushu G. Cancellous bone block allografts for the augmentation of the anterior atrophic maxilla. Clin Implant Dent Relat Res. 2011 Jun;13(2):104-11. doi: 10.1111/j.1708-8208.2009.00193.x. PMID 19744202